CLINICAL TRIAL: NCT01801657
Title: The Role of Viral Infection in Acute Exacerbations of Non-cystic Fibrosis Bronchiectasis in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, yonghua gao, PHD, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 2009CB522109
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; exacerbation; virus
MeSH Terms: conditions — Bronchiectasis; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bronchiectasis,stable: A patient was defined as stable if there was no exacerbation for the previous 4 wk
- Bronchiectasis,exacerbations: Bronchiectasis exacerbations were defined by subjective and persistent(>24 h) deterioration in at least three respiratory symptoms, including cough, dyspnea, hemoptysis, increased sputum purulence or volume, chest pain (with or without fever), radiographic deterioration, systemic disturbances, or changes in chest auscultation

SUMMARY:
Bronchiectasis is clinically characterized by irreversible dilation of the bronchi and bronchioles leading to persistent cough, purulent sputum, and airway ﬂow limitation, which may be accompanied by recurrent exacerbations.It has been increasingly recognized that respiratory viruses are mainly responsible for acute exacerbation of chronic pulmonary diseases, i.e. asthma, chronic obstructive pulmonary disease and cystic fibrosis. However,little is known about the roles of viral infection in driving exacerbations of bronchiectasis.This study aims to identify the frequency of common viral infections and determine the roles that viruses play in acute exacerbations of bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic airway disease characterised by a vicious cycle of persistent bacterial colonization,inflammation and progressive tissue destruction.Patients with bronchiectasis frequently developed acute exacerbations characterised by acute worsening requiring changes in concomitant use of medication,with attendant adverse effects on their morbidity and health-related quality of life. The detailed pathogenesis of exacerbations of bronchiectasis, however, remains poorly understood.

Recent data suggested that airway infection and inflammation are important drivers of exacerbations,therefore the imbalance between chronic bacterial infection and host immune response may result in bronchiectasis exacerbations. Viral infection may be an important factor that leads to this events.It has been established that respiratory viruses are mainly responsible for the exacerbations of other chronic respiratory diseases, i.e. asthma, COPD and cystic fibosis. However, the data regarding prospective studies that sought to investigate the roles of viruses in acute exacerbation of bronchiectasis are lacking. Furthermore,the associations between viruses and bacteria during exacerbation need to be assessed. This study targets at indentifying the frenquency of common viral infections in adults with non-cystic fibrosis bronchiectasis and may shed light on the effects they have on clinical parameters,i.e. the length of exacerbated symptom to recovery,lung function, pulmonary inflammation, bacterial load and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HRCT-diagnosed Bronchiectasis
* Capable of providing written informed consent

Exclusion Criteria:

* Patient judged to have poor compliance
* Cystic fibrosis bronchiectasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with non-CF bronchiectasis diagnosed by High Resolution CT(HRCT) attending the out-patient clinics of First Affiliated Hospital of Guangzhou Medical University,Guangzhou,Guangdong,China
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The prevalence of respiratory virus infection in adults with bronchiectasis during a pulmonary exacerbation and when clinically stable. | 1 year
  Respiratory viruses in the nasal swab and sputum will be identified using the polymerase chain reaction(PCR)technique when clinically stable and during exacerbation.The following viruses will be tested for:influenza A,B(including influenza A H1N1),respiratory syncytial virus(RSV),Enterovirus,Parainfluenza 1-4,Rhinovirus,human Coronaviruses(subtypes OC43、229E、HKU1),human metapneumovirus,adenovirus, human bocavirus,chlamydia,mycoplasma.

SECONDARY OUTCOMES:
The effect of respiratory virus infection on systemic and pulmonary inflammatory markers. | 1 year
  Systemic and airway inflammatory cytokines including IL-1β、IL-6、IL-8、TNF-a were measured using a commercial multiplex bead-based assay.
The effect of respiratory virus on lung function | 1 year
  Spirometric indices in the present study is referred to as forced expiratory vilume in 1s(FEV1),forced vital capacity(FVC).Spirometry tests are carried out using a spirometer (COSMED, QUARK PFT, Italy). All operation procedures meet the joint recommendation by ATS and ERS. A total of at least 3 (not more than 8) spirometric maneuvers are performed, with the variation between the best two maneuvers of <5% or 200ml in FVC and FEV1. The maximal values of FVC and FEV1 are reported.
The effect of respiratory virus infection on the bacterial load in bronchiectasis. | 1 year
  Type of bacterial infection, also referred to as potentially pathogenic organisms, and bacterial load, as expressed in cfu per mililiter
Time to recovery of respective symptom | 1 year
  The time from exacerbation onset by which a 3-d moving average was equal to or exceeded the baseline value
The effect of respiratory virus on quality of life in patients with bronchiectasis | 1 year
  Quality of life in patients with bronchiectasis were measured by St.George Respiratory Questionnaire、Leicester Cough Questionnaire and COPD assessment test during exacerbations,and then compared between virus-postive and virus-negative patients
To investigate if upper respiratory tract symptoms are associated with viral infections. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Nanshan Zhong, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Gao YH, Guan WJ, Xu G, Lin ZY, Tang Y, Lin ZM, Gao Y, Li HM, Zhong NS, Zhang GJ, Chen RC. The role of viral infection in pulmonary exacerbations of bronchiectasis in adults: a prospective study. Chest. 2015 Jun;147(6):1635-1643. doi: 10.1378/chest.14-1961. PMID 25412225